CLINICAL TRIAL: NCT00314795
Title: An Open-Label Study to Investigate the Efficacy and Safety of AF37702 Injection in the Treatment of Anemia Caused by Antibody-Mediated Pure Red Cell Aplasia in Patients With Chronic Kidney Disease
Brief Title: Efficacy and Safety of Peginesatide (AF37702) in the Treatment of Anemia in Participants With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-06; 2005-004944-30 (EudraCT Number)
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Anemia; Chronic Kidney Disease; Chronic Renal Failure; Pure Red Cell Aplasia
Keywords: Drug Therapy; pure red cell aplasia; PRCA; chronic kidney disease; CKD; chronic renal failure; CRF; anemia; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; hemoglobin; Hb; Hgb; red blood cell; red blood cell production
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Red-Cell Aplasia, Pure | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peginesatide (Experimental): Peginesatide 0.05 mg/kg injection, subcutaneously as a starting dose followed by peginesatide 0.1 mg/kg injection, subcutaneously once every 4 weeks for up to 6 months.
  Individual dose of peginesatide injection was modified based on hemoglobin levels. Dose adjustments were made in order to achieve and maintain hemoglobin in the target range of 10.0-12.0 g/dL.
  Interventions: Drug: Peginesatide

INTERVENTIONS:
Drug: Peginesatide — Peginesatide injection
  Other Names: Omontys; Hematide; AF37702

SUMMARY:
The purpose of this study is to evaluate the ability of peginesatide (AF37702) to increase and maintain increased hemoglobin levels in participants with chronic kidney disease (CKD) (either not on dialysis, receiving regular hemodialysis or peritoneal dialysis, or following renal transplant) with confirmed antibody-mediated pure red cell aplasia (PRCA).

DETAILED DESCRIPTION:
The drug being tested in this study was peginesatide. Peginesatide injection was tested to investigate the efficacy and safety in the treatment of anemia caused by antibody-mediated pure red cell aplasia in participants with chronic kidney disease.

The study enrolled 22 patients. All the participants enrolled into the study received:

• Peginesatide 0.5 mg/kg subcutaneous (SC) injection

The participants received a starting dose of 0.05 mg/kg (every 4 weeks) followed by 0.1 mg/kg dose, based on the assessment of the dose response in the initial group of 5 participants. The frequency of each injection and the dose adjusted based on the participant's hemoglobin response and the ability to maintain a hemoglobin level in the range of 10.0-12.0 g/dL.

This multi-center trial was conducted in Europe. The overall time to participate in this study was 10 years and 7 months approximately. Participants made multiple visits to the clinic until the projected end of treatment period, which was 31-Oct-2016.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have confirmed antibody-mediated Pure red cell aplasia (PRCA) are potentially eligible for enrollment into this study.
* Participants must be ≥ 18 years old at the time of consent.
* Erythropoiesis stimulating agents (ESAs) must be discontinued for a minimum of 1 month prior to screening.
* Participant requires periodic transfusions to maintain hemoglobin.
* Hemoglobin < 10 g/dL for at least 2 measurements or participant has received a transfusion within the past 4 weeks to achieve a hemoglobin > 10 g/dL.
* Confirmation that an anti-erythropoietin antibody sample was obtained for analysis by the central reference laboratory within 1 month prior to baseline.
* Participants can either be participants with chronic kidney disease not yet requiring renal replacement therapy (participants not on dialysis), those on regular hemodialysis or peritoneal dialysis, or following a renal transplant.
* Participants may or may not have previously been treated with immunosuppressive therapy.
* Pre-menopausal females (with the exception of those who are surgically sterile) must have a negative pregnancy test at screening.
* Written informed consent must be obtained.

Exclusion Criteria:

* Participants already successfully on another erythropoietic agent.
* Abnormal bone marrow findings consistent with the diagnosis of myelodysplasia, a myeloproliferative disorder, hematologic malignancy or evidence of metastatic infiltration.
* Poorly controlled hypertension.
* Previous exposure to any investigational agent within 4 weeks prior to administration of study drug or planned receipt during the study period.
* High likelihood of early withdrawal or interruption of the study.
* Participants who refuse to give informed consent.
* Women who are pregnant, lactating or not using a medically approved birth control.
* Life expectancy <12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-04-06 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (4):
- Research Facility, Paris, France
- Research Facility, Erlangen, Germany
- United Kingdom (2):
  - Research Facility, Derby
  - Research Facility, London

REFERENCES:
- [Result] Macdougall IC, Rossert J, Casadevall N, Stead RB, Duliege AM, Froissart M, Eckardt KU. A peptide-based erythropoietin-receptor agonist for pure red-cell aplasia. N Engl J Med. 2009 Nov 5;361(19):1848-55. doi: 10.1056/NEJMoa074037. PMID 19890127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Europe from 06-Apr-2006 to 31-Oct-2016.
Pre-assignment Details: Participants with a diagnosis of chronic renal failure (CRF) with confirmed antibody-mediated pure red cell aplasia (PRCA) were enrolled to receive peginesatide subcutaneous injection up to 0.3 mg/kg, once every 4 weeks for up to 60 months.
Groups:
- Peginesatide: Peginesatide 0.05 mg/kg injection, subcutaneously followed by peginesatide 0.1 mg/kg injection, subcutaneously once every 4 weeks for up to 60 months.
  Individual dose of peginesatide injection was modified based on hemoglobin levels. Dose adjustments were made in order to achieve and maintain hemoglobin in the target range of 10.0-12.0 g/dL.
Period: Overall Study
Arm/Group | Peginesatide
Started | 22
Completed | 2
Not Completed | 20
Not completed — Adverse Event | 8
Not completed — Death | 4
Not completed — Reason not Specified | 3
Not completed — Renal Transplant | 3
Not completed — Participants Withdrew Consent | 2

BASELINE CHARACTERISTICS:
Population: Full analysis population is defined as all participants enrolled and started on study treatment.
Arm/Group | Peginesatide
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  Caucasian | 17
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  France | 6
  Germany | 8
  United Kingdom | 8
Height [Mean (Standard Deviation); unit: cm] — Population: Here, number analyzed are the participants who were evaluated for this baseline measure.
  cm
    number analyzed (Participants) | 21
    (all) | 168.1 (9.66)
Weight [Mean (Standard Deviation); unit: kg] | 67.6 (12.31)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Here, number analyzed are the participants who were evaluated for this baseline measure.
  kg/m^2
    number analyzed (Participants) | 21
    (all) | 23.8 (2.41)
Baseline Hemoglobin (Hgb) [Mean (Standard Deviation); unit: g/L] | 96.5 (16.11)
Baseline Ferritin [Mean (Standard Deviation); unit: ug/L] — Population: Here, number analyzed are the participants who were evaluated for this baseline measure.
  ug/L
    number analyzed (Participants) | 21
    (all) | 2332.0 (1695.02)
Baseline Transferrin Saturation [Mean (Standard Deviation); unit: % transferrin] — Population: Here, number analyzed are the participants who were evaluated for this baseline measure.
  % transferrin
    number analyzed (Participants) | 19
    (all) | 79.2 (21.87)
Baseline Anti-erythropoietin (EPO) Antibody Titers [Mean (Standard Deviation); unit: U/mL] | 94.1 (217.08)
Bone Marrow Evaluation [Count of Participants; unit: Participants] — Here Erythroblastopenia=EBP; Hypoplasia= HYP; Hypocellular=hpc; bone marrow=BM; Erythroid lineage-EL; diagnosis=dgn; reticulocyte=retic.
  Participants
    Aplasia of Erythropoese | 1
    Erythroblastopenia (EBP) | 1
    EBP 0% normal values for other cell lineages | 1
    Erythroid series absent | 1
    Erythroid severe HYP no decrease in other lineages | 1
    Erythropoietic hypoplasia | 1
    Hpc BM with reduced EL consistent with dgn of pure | 1
    HYP of erythropoiesis staining of iron in BM retic | 1
    Normal | 1
    PRCA | 8
    PRCA / Bone Marrow Trephine | 1
    Pure Red Cell Aplasia | 2
    Red cell aplasia | 1
    Red cell hypoplasia | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Increase and Maintain Hemoglobin Levels (Two Consecutive Values) Greater Than or Equal to the Lower Limit of the Target Range in the Absence of Red Blood Cell Transfusion in the Previous 28 Days by Week 24
Description: Percentage of participants who experienced increase and maintain hemoglobin levels (two consecutive values) greater than or equal to the lower limit (11 g/dL) in the absence of red blood cell transfusion in the previous 28 days by week 24 were reported.
Time Frame: Up to Week 24
Population: Efficacy endpoint data was not collected due to low patient enrollment and the drug was withdrawn from the market.
Arm/Group | Peginesatide
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Red Blood Cells (RBCs) Transfusions During the 26 Weeks Pre-treatment Period (Prior to Enrollment) and During 13- and 26 Weeks Intervals During the Study
Time Frame: 26 weeks prior to enrollment up to end of study (up to 60 months)
Population: Efficacy endpoint data was not collected due to low patient enrollment and the drug was withdrawn from the market.
Arm/Group | Peginesatide
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With RBC Transfusions During the 26-week Pre-treatment Period and During 13- and 26-week Intervals During the Study
Time Frame: 26 weeks prior to enrollment up to end of study (up to 60 months)
Population: Efficacy endpoint data was not collected due to low patient enrollment and the drug was withdrawn from the market.
Arm/Group | Peginesatide
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Initial Achievement of Hemoglobin (Hgb) Greater Than or Equal to the Lower Limit of the Target Range in the Absence of Red Blood Cell Transfusions in the Previous 28 Days
Description: The time between first dose administered and the initial achievement of a Hgb increase ≥11 g/dL for two consecutive visits was calculated for each participant as the number of days between the first dose administration date and the earlier of (1) the study termination date [i.e. censor date] and (2) the first date of an Hgb increase ≥ 11 g/dL for two consecutive visits without whole blood or RBC transfusion during the previous 28 days. Time to initial Hgb increase ≥ 11 g/dL will be calculated for each participant as the minimum of censor date and increase date minus the first dose date plus 1.
Time Frame: Up to 60 months
Population: Efficacy endpoint data was not collected due to low patient enrollment and the drug was withdrawn from the market.
Arm/Group | Peginesatide
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Leading to Treatment Discontinuation
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From signing of informed consent form up to Month 60
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Peginesatide
Number analyzed (Participants) | 22
Participants
  AEs | 22
  SAEs | 17
  AEs Leading to Study Drug Discontinuation | 3

ADVERSE EVENTS:
Time Frame: From signing of informed consent form up to Month 60
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Peginesatide
Serious Adverse Events (participants affected / at risk) | 17/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=22)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2 — One treatment-emergent death occurred and is not related to the study drug.
Cardiac failure (Cardiac disorders) | 3 — One treatment-emergent death occurred and is not related to the study drug.
Cardiac failure acute (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Optic ischaemic neuropathy (Eye disorders) | 1
Anal prolapse (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 — One treatment-emergent death occurred and is not related to the study drug.
Chest Pain (General disorders) | 1
Death (General disorders) | 1 — Treatment-emergent death is not related to the study drug.
Sudden death (General disorders) | 1 — Treatment-emergent death is not related to the study drug.
Vascular stent restenosis (General disorders) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Disseminated tuberculosis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1 — One treatment-emergent death occurred and is not related to the study drug.
Urosepsis (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
C-reactive protein increased (Investigations) | 1
Drug specific antibody present (Investigations) | 1
Haematocrit decreased (Investigations) | 1 — One treatment-emergent death occurred and is not related to the study drug.
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — One treatment emergent death occurred and is related to the study drug.
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vascular dementia (Nervous system disorders) | 1
Renal salt-wasting syndrome (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 — One treatment-emergent death occurred and is not related to the study drug.
Aortic stenosis (Vascular disorders) | 1
Blood pressure inadequately controlled (Vascular disorders) | 1
Femoral artery aneurysm (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=22)
Palpitations (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Cataract (Eye disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 3
Vomitting (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Oedema peripheral (General disorders) | 7
Asthenia (General disorders) | 6
Fatigue (General disorders) | 5
Non-cardiac chest pain (General disorders) | 2
Pyrexia (General disorders) | 2
Hepatomegaly (Hepatobiliary disorders) | 2
Drug hypersensitivity (Immune system disorders) | 3
Seasonal allergy (Immune system disorders) | 2
Nasopharyngitis (Infections and infestations) | 10
Bronchitis (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 3
Cystitis (Infections and infestations) | 2
Cytomegalovirus infection (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 8
Skin abrasion (Injury, poisoning and procedural complications) | 5
Contusion (Injury, poisoning and procedural complications) | 2
Heat exhaustion (Injury, poisoning and procedural complications) | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 2
Haemoglobin decreased (Investigations) | 6
Weight decreased (Investigations) | 4
Blood pressure increased (Investigations) | 3
Blood phosphorus increased (Investigations) | 2
Blood potassium increased (Investigations) | 2
Liver function test increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Reticulocyte count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 4
Fluid overload (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscke spasms (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Restless legs syndrome (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Haematuria (Renal and urinary disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 4
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 6
Haematoma (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.